CLINICAL TRIAL: NCT01905462
Title: Post-marketing Safety Study to Assess the Risk of Spontaneous Abortions in Women Exposed to Cervarix in the United Kingdom
Brief Title: Post-marketing Safety Study to Assess the Risk of Spontaneous Abortions in Women Exposed to Cervarix Residing in UK
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Clinical Practice Research Datalink (Other Government)
Responsible Party: Sponsor
Other Study IDs: 114101
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Infections, Papillomavirus
Keywords: Cervarix; Spontaneous abortion; Vaccine; Human Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections; Abortion, Spontaneous | interventions — Data Collection; human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed cohort: Women with the first day of LMP between 30 days before and 45 days after any Cervarix dose and between 30 days before and 90 days after any Cervarix dose.
  Interventions: Other: Data Collection; Biological: Cervarix
- Non-exposed cohort: Women with the first day of LMP between 120 days and 18 months after their last Cervarix dose (and no further Cervarix dose before the outcome).
  Interventions: Other: Data Collection; Biological: Cervarix

INTERVENTIONS:
Other: Data Collection — Analyses of data collected within the CPRD GOLD database.
Biological: Cervarix — Women with last menstrual period (LMP) between 30 days before and 45 days after, or 30 days before and 90 days after any dose of Cervarix and women with LMP between 120 days and 18 months after the last Cervarix dose.

SUMMARY:
This study will assess the risk of spontaneous abortion during weeks 1-23 and weeks 1-19 of gestation, respectively, and other pregnancy outcomes, in an exposed cohort, i.e. women with last menstrual period (LMP) between 30 days before and 45 days after, or 30 days before and 90 days after any dose of Cervarix, when compared to a non-exposed cohort, i.e. women with LMP between 120 days and 18 months after the last Cervarix dose. The data collected in the Clinical Practice Research Datalink General Practitioner OnLine Database (CPRD GOLD) in the UK, will be analysed in this study.

DETAILED DESCRIPTION:
Convenience sampling will be used in this study. It is planned to include all eligible pregnant women (included in CPRD GOLD and who fulfil to the inclusion/exclusion criteria) in each of the two cohorts.

ELIGIBILITY:
Inclusion Criteria:

For the exposed cohort:

All subjects must satisfy all of the following criteria at entry into the exposed cohort:

* Full date of first day of LMP available in the database or calculated from Estimated date of delivery (EDD).
* Female, aged between, and including, 15 and 25 years of age at LMP.
* Recorded in the CPRD GOLD for at least 12 months at LMP.
* First day of LMP available in the database or calculated from EDD between September 1st 2008 and June 30th 2011.
* At least one dose of Cervarix received between September 1st 2008 and June 30th 2011.
* Full date of Cervarix vaccination(s) available.
* First day of LMP available in the database or calculated from EDD between 30 days before and 90 days after any dose of Cervarix.
* Subject defined as acceptable in CPRD GOLD.

For the non-exposed cohort:

All subjects must satisfy all of the following criteria at entry into the non-exposed cohort:

* Full date of first day of LMP available in the database or calculated from EDD.
* Female, aged between, and including, 15 and 25 years of age at LMP.
* Recorded in the CPRD GOLD since at least 12 months at LMP.
* First day of LMP available in the database or calculated from EDD between September 1st 2008 and June 30th 2011.
* At least one dose of Cervarix received between September 1st 2008 and June 30th 2011.
* Full date of Cervarix vaccination(s) available.
* First day of LMP available in the database or calculated from EDD between 120 days and 18 months after the last dose of Cervarix.
* Subject defined as acceptable in CPRD GOLD.

Exclusion Criteria:

For the exposed cohort:

• Female with the first day LMP between 30 days before and 90 days after at least one dose of unspecified Human Papillomavirus vaccine and/or Gardasil.

For the non-exposed cohort:

* Female with the first day LMP between 30 days before and 90 days after at least one dose of unspecified Human Papillomavirus vaccine and/or Gardasil.
* Female included for a previous pregnancy in the exposed cohort.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women aged 15 to 25 years, residing in UK, exposed to Cervarix and whose data is recorded in the CPRD GOLD.
Sampling Method: Non-Probability Sample
Enrollment: 1046 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of spontaneous abortion | Weeks 1-23 of gestation

SECONDARY OUTCOMES:
Occurrence of spontaneous abortion | Weeks 1-19 of gestation
Occurrence of other pregnancy outcomes | 12 months after last menstrual period
  Induced/therapeutic and other abortions; Stillbirth; Birth defects identified among all pregnancies with known outcome classified as live births, stillbirths and abortions. For live births, birth defects identified within the first 12 weeks of life will be included; Small/large for gestational age at birth; Pre-term and post-term delivery.
Baby's death | First 12 weeks of baby's life

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom